CLINICAL TRIAL: NCT06850805
Title: A 12-Week Randomized, Double-Blind, Placebo-Controlled, Multicenter Study Evaluating the Efficacy and Safety of Intranasal Administration of 186 mcg of OPN-375 Twice a Day (BID) in Adolescent Subjects With Chronic Rhinosinusitis Without Nasal Polyps
Brief Title: Efficacy and Safety of 186 mcg of OPN-375 Nasal Spray Twice a Day (BID) in Adolescents With Chronic Rhinosinusitis Without Nasal Polyps
Acronym: Re-Open 3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Optinose US Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPN-FLU-CS-3207
Record Dates: First submitted 2025-02-14; First posted 2025-02-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Chronic Rhinosinusitis Without Nasal Polyps
Keywords: Chronic Sinusitis; Chronic Rhinosinusitis; XHANCE

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo BID (Placebo Comparator): Double-Blind Treatment Phase: Intranasal administration of matching placebo BID x 12 weeks
  Interventions: Drug: Placebo
- OPN-375 186 µg BID (Active Comparator): Double-Blind Treatment Phase: Intranasal administration of OPN-375 186 µg x 12 weeks
  Interventions: Drug: OPN-375

INTERVENTIONS:
Drug: OPN-375 — OPN-375 (fluticasone propionate) delivered via exhalation delivery system (EDS) BID
  Arms: OPN-375 186 µg BID
Drug: Placebo — Placebo solution administered via exhalation delivery system (EDS).
  Arms: Placebo BID

SUMMARY:
This is a 12-Week randomized, double-blind, placebo-controlled, parallel-group, multicenter study evaluating the efficacy and safety of intranasal administration of 186 µg of OPN-375 twice a day (BID) in adolescent subjects with chronic rhinosinusitis without nasal polyps. The total planned number of subjects is approximately 84 adolescents (12-17 years of age) who will be randomly assigned to receive 1 of 2 study treatments using a 1:1 ratio (OPN-375 186 µg:placebo). The study includes a PK sub-study, in which up 14 subjects will be enrolled to obtain 10 completers.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the efficacy of intranasal administration of OPN-375 (fluticasone propionate)186 µg twice a day (BID) versus placebo in adolescents with chronic rhinosinusitis (CRS) without nasal polyps (sNP) using the endpoint of change from baseline in CRS symptoms as measured by a 7-day average instantaneous composite score of nasal symptoms (CSS) at the end of Week 4. The CSS is the sum of scores assigned to the symptoms congestion, facial pain or pressure sensation, and nasal discharge (anterior and/or posterior), on a scale of 0 (non-symptomatic) to 3 (severe symptoms). The total CSS can range from 0-9. Eligible study subjects will complete a 7 to 21 day screening period followed by a 12-week double-blind treatment period, for a total of approximately 15 weeks of participation. The study consists of 3 on-site study visits (screening/V1, randomization/V2, end of study/V3/Week 12) and two telephone calls at participation weeks 4 and 8.

The study will include a pharmacokinetic (PK) substudy in which PK assessment of 186 µg OPN-375 in up to 14 study subjects will be conducted in an open label fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 12 to 17 years, inclusive, at time of Visit 1 (Screening)
2. Female subjects, if sexually active, must:

   1. be practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method [e.g., condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel], or male partner sterilization) before entry and throughout the study, or
   2. be surgically sterile, (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy), or
   3. be abstinent.
3. Females of child-bearing potential must have a negative urine pregnancy test at Visit 1 (Screening).
4. Must have a history of CRS and be currently experiencing 2 or more of the following symptoms, 1 of which has to be either nasal congestion or nasal discharge (anterior and/or posterior nasal discharge) for equal to or greater than 12 weeks:

   * nasal congestion
   * nasal discharge (anterior and/or posterior nasal discharge)
   * facial pain or pressure
   * reduction or loss of smell
5. Must have endoscopic evidence of nasal mucosal disease, with edema, or purulent discharge bilaterally, or presence of bilateral disease on a prior computed tomography (CT) scan performed within 14 days of Visit 1.
6. Must have at least moderate symptoms (as defined in protocol) of nasal congestion as reported by the subject, on average, for the 7-day period preceding Visit 1 (Screening) run-in.
7. Must have an average morning score of at least 1.5 for congestion on the Nasal Symptom Scale (as defined in protocol) recorded on the subject diary over a 7-day period during the first 14 days of the single-blind run-in period.
8. Must demonstrate an ability to correctly complete the daily diary during the run-in period to be eligible for randomization.
9. Subjects with comorbid asthma must be stable, defined as no exacerbations (e.g., no emergency room visits, hospitalization, or oral or parenteral steroid use) within the 3 months before Visit 1 (Screening). Subjects who received inhaled corticosteroids are required to be on no more than a moderate dosage regimen as defined by 2021 Global Initiative for Asthma Guidelines (GINA) for 1 month before Visit 1 (Screening), and are expected to remain on it throughout the study. Subjects receiving inhaled fluticasone alone or in combination may not participate in the PK sub-study.
10. Subjects with aspirin exacerbated respiratory disease, who have undergone aspirin desensitization and are receiving daily aspirin therapy, must be receiving therapy for at least 6 months prior to Visit 1.
11. Must be able to cease treatment with intranasal steroids, inhaled corticosteroids (except permitted doses listed above for asthma) at the screening visit
12. If taking oral antihistamines, must be on a stable regimen for at least 2 weeks prior to Visit 1 (Screening), and agree to not change the dose of these medications until after Week 4 of the study.
13. Must be able to use the exhalation delivery system (EDS) correctly; all subjects will be required to demonstrate correct use with the practice EDS at Visit 1 (Screening).
14. Must be capable, in the opinion of the investigator, of providing assent and parent or guardian must provide informed consent to participate in the study. Subjects must sign an informed consent document indicating that they understand the purpose of and procedures required for the study and that they are willing to participate in the study.

Exclusion Criteria:

1. Females who are pregnant or lactating.
2. Inability to have each nasal cavity examined for any reason, including nasal septum deviation.
3. Inability to achieve bilateral nasal airflow.
4. Is currently taking XHANCE®.
5. Have previously used XHANCE for more than 1 month and did not achieve an adequate symptomatic response.
6. History of sinus or nasal surgery within 6 months before Visit 1 or has not healed from a prior sinus or nasal surgery.
7. Have current evidence of odontogenic sinusitis, sinus mucocele (the affected sinus is completely opacified and either the margins are expanded and/or thinned OR there are areas of complete bone resorption resulting in bony defect and extension of the "mass" into adjacent tissues), evidence of allergic fungal sinusitis, or evidence of complicated sinus disease (including, but not limited to, extension of inflammation outside of the sinuses and nasal cavity).
8. Have a paranasal sinus or nasal tumor.
9. Have a nasal polyp score of grade 1 or greater in either nostril as determined by the nasoendoscopy at screening.
10. Have a nasal septum perforation.
11. Have had more than 1 episode of epistaxis with frank bleeding in the month before Visit 1 (Screening).
12. Have evidence of significant mucosal injury, ulceration (eg, exposed cartilage) on Visit 1 (Screening) nasal examination/nasoendoscopy.
13. Have current, ongoing rhinitis medicamentosa (rebound rhinitis).
14. Have significant oral structural abnormalities (eg, a cleft palate).
15. Have a diagnosis of cystic fibrosis.
16. History of eosinophilic granulomatosis with polyangiitis (Churg-Strauss syndrome).
17. Symptom resolution or last dose of antibiotics for purulent nasal infection, acute sinusitis, or upper respiratory tract infection, influenza, or SARS-CoV-2 (COVID-19) has not occurred before Visit 1. Potential subjects presenting with any of these infections may be rescreened 4 weeks after symptom resolution.
18. Planned sinonasal surgery during the period of the study.
19. Allergy, hypersensitivity, or contraindication to corticosteroids or steroids.
20. Has used oral steroids in the past for treatment of CS and did not experience any relief of symptoms.
21. Has a steroid eluting sinus stent still in place within 30 days of Visit 1.
22. Allergy or hypersensitivity to any excipients in study drug.
23. Exposure to any glucocorticoid treatment with potential for systemic effects (eg, oral, parenteral) within 1 month before Visit 1 (Screening); except as noted in inclusion criteria for subjects with comorbid asthma or COPD.
24. Have nasal or oral candidiasis.
25. History or current diagnosis of any form of glaucoma or ocular hypertension.
26. History of IOP elevation on any form of steroid therapy.
27. History or current diagnosis of the presence (in either eye) of a cataract unless both natural intraocular lenses have been removed.
28. History of immunodeficiency of any etiology (including poor nutrition) that would be anticipated to affect the likelihood of benefit or harm from the therapeutic intervention.
29. Any serious or unstable concurrent disease, psychiatric disorder, or any significant condition that, in the opinion of the investigator could confound the results of the study or could interfere with the subject's participation or compliance in the study.
30. Have a positive drug screen or a history of drug or alcohol abuse, or dependence that, in the opinion of the investigator could interfere with the subject's participation or compliance in the study.
31. Have participated in an investigational drug clinical trial within 30 days of Visit 1 (Screening).
32. Have received mepolizumab (Nucala®), reslizumab (Cinquair®), dupilumab (Dupixent®), omalizumab (Xolair®), benralizumab (Fasenra™), Tezepelumab-ekko (Tezspire®) or any other immune-modifying monoclonal antibody within 6 months of Visit 1 (Screening).
33. Is using strong cytochrome P450 3A4 (CYP3A4) inhibitor (eg, ritonavir, atazanavir, clarithromycin, indinavir, itraconazole, nefazodone, nelfinavir, saquinavir, ketoconazole, telithromycin, conivaptan, lopinavir, voriconazole, cobicistat).
34. Has a parent, guardian or caregiver who is an employee of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, or is a family member of the employee or the investigator.
35. Patients who report unexplained worsening of vision within the past 3 months.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to the end of Week 4 in the average instantaneous CSS (evaluation of symptom severity immediately preceding the time of scoring). | 4 Weeks
  The CSS consists of the sum of the scores (0-3) assigned to each of the following symptoms of CRS: nasal congestion, nasal discharge (anterior and/or posterior), facial pain/pressure sensation, where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, and 3 = severe symptoms. The total CSS for each day can range from 0 to 9. Participants will report symptom severity immediately preceding the time of scoring every morning (AM). The baseline CSS is the average of the CSS's over the last 7 days of the single-blind run-in period. The end of Week 4 CSS is the average of the CSS's over the 7 days before Week 4.

SECONDARY OUTCOMES:
Frequency of acute exacerbations of CRS over the 12-week treatment period | 12 weeks
  Acute exacerbations of CRS (AECRS) are defined as a worsening of symptoms that requires an escalation of treatment. The number of AECRS experienced by each participant will be recorded.
Change from baseline to the end of Week 4 on CSS score in subjects using an intranasal steroid treatment for CRS within 30 days of Visit 1/Screening | 4 Weeks
  The CSS consists of the sum of the scores (0-3) assigned to each of the following symptoms of CRS: nasal congestion, nasal discharge (anterior and/or posterior), facial pain/pressure sensation, where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, and 3 = severe symptoms. The total CSS for each day can range from 0 to 9. Participants will report symptom severity immediately preceding the time of scoring every morning (AM). The baseline CSS is the average of the CSS's over the last 7 days of the single-blind run-in period. The end of Week 4 CSS is the average of the CSS's over the 7 days before Week 4. This outcome will assess this change in CSS specifically in the subgroup of participants who were symptomatic at trial entry despite reported use of an intranasal steroid for treatment of CRS within 30 days of Visit 1/Screening.
Change from baseline to the end of Weeks 8 and 12 in CSS | 8 Weeks; 12 Weeks
  The CSS consists of the sum of the scores (0-3) assigned to each of the following symptoms of CRS: nasal congestion, nasal discharge (anterior and/or posterior), facial pain/pressure sensation, where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, and 3 = severe symptoms. The total CSS for each day can range from 0 to 9. Participants will report symptom severity immediately preceding the time of scoring every morning (AM). The baseline CSS is the average of the CSS's over the last 7 days of the single-blind run-in period. The CSS for the end of Week 8 and Week 12 is the average of the CSS's over the 7 days before Week 8 and Week 12, respectively.
Change from baseline to the end of Weeks 4, 8 and 12 in four separate cardinal CRS symptoms | 4 Weeks; 8 Weeks; 12 Weeks
  Participants will rate each of the following four cardinal symptoms of CRS every morning based on symptom severity immediately before reporting: nasal congestion, facial pain or pressure sensation, nasal discharge (anterior and/or posterior), and sense of smell. Participants will rate each symptom on a scale of 0 to 3, where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, and 3 = severe symptoms. Scores from the 7 days immediately preceding each timepoint will be averaged. The change in 7-day average score from baseline to Week 4, Week 8, and Week 12 for each symptom will be assessed individually.
Percent of subjects indicating improvement on the Patient Global Impression of Change (PGIC) at Week 12/ end of study. | 12 Weeks
  The Patient Global Impression of Change (PGIC) survey consists of a single question asking participants to rate how much their symptoms have changed since beginning use of the study drug on a scale of 1 to 7, where 1 = Very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. The percent of subjects indicating any improvement (minimal, much, or very much) will be assessed.
Change from baseline to Week 12 in the 5 domains of the SN-5 Questionnaire | 12 Weeks
  The SN-5 questionnaire is a quality of life assessment that will be completed by the participant/parent. There are 5 specific symptom related questions (answered on a 7-point Likert scale on frequency of symptoms, where 1 = none of the time and 7 = all of the time), and 1 general quality of life question, answered on a visual analog scale from 0 (worst) to 10 (best). For this outcome, the change in score from baseline to Week 12/end of participation will be assessed for each of the 5 symptom related questions.
Change from baseline to Week 12 in overall quality of life as measured by the SN-5 Questionnaire | 12 Weeks
  The SN-5 questionnaire is a quality of life assessment that will be completed by the participant/parent. There are 5 specific symptom related questions (answered on a 7-point Likert scale on frequency of symptoms, where 1 = none of the time and 7 = all of the time), and 1 general quality of life question, answered on a visual analog scale from 0 (worst) to 10 (best). This outcome will assess the change in score from baseline to Week 12/end of participation for general quality of life question.

OTHER OUTCOMES:
Assessment of safety through Adverse Events (AEs) | 12 Weeks
  Safety will be assessed by reporting frequency and severity (mild, moderate, or severe) of AEs experienced by participants during the trial. AEs will be collected beginning at time of signing of the Informed Consent Form (ICF) through end of participation (Week 12 or early termination).
Assessment of safety by nasal examination | 12 Weeks
  Nasal examinations will be completed on all participants via nasoendoscopy at screening and end of study (Week 12 or early termination). Physicians performing the nasoendoscopies will record the presence of epistaxis, septal erosion/perforation, and details related to ulceration/erosion of any area other than the septum. The frequency and severity of findings from these exams will be reported.
Assessment of safety by ocular examination visual acuity | 12 Weeks
  Ocular examinations will be performed during screening period and end of participation (Week 12 or early termination), and will include an assessment of visual acuity. Visual acuity will be assessed using an eye chart (EVA, EDTRS or Snellen) and will be recorded for each eye in the form of a fraction: 20/x.
Assessment of safety by ocular examination intraocular pressure (IOP) | 12 Weeks
  Ocular examinations will be performed during screening period and end of participation (Week 12 or early termination), and will include an assessment of intraocular pressure. Intraocular pressure will be assessed using a Goldmann applanation tonometer mounted on a slit lamp, a hand-held applanation Goldmann-type tonometer, or a Tono-Pen. Two measurements will be performed for each eye. If the first 2 measurements differ by more than 3 mm Hg, a third measurement will be performed. The average value of the 2 or 3 measurements will be calculated. Subjects in whom IOP is elevated above 21 mm Hg will not be enrolled. Any new occurrence of intraocular pressure elevation above 21 mm Hg will require subject withdrawal.
Assessment of safety by ocular examination for cataracts | 12 Weeks
  Ocular examinations will be performed during screening period and end of participation (Week 12 or early termination), and will include an assessment of presence of cataracts. Each of the participant's eyes will be assessed for the presence of cataracts. If a cataract is identified, it will be specified based on type (nuclear, cortical, or posterior subcapsular) and assigned a grade of 1, 1+, 2, 2+, 3, 3+, or 4. Participants with cataracts at screening will not be enrolled. Any new occurrence of cataracts of any grade will require withdrawal from the study.
Assessment of safety by weight measurement | 12 Weeks
  Participant weight will be collected at screening, randomization and end of participation (Week 12 or early termination). Weight will be measured in kilograms or pounds and findings will be summarized using descriptive statistics including mean values and change from baseline values, as well as numbers of subjects with values outside limits of the normal range at each time point.
Assessment of safety by measuring vital signs - blood pressure | 12 Weeks
  Participant blood pressure measurements will be collected at screening, randomization and end of participation (Week 12 or early termination). Systolic and diastolic blood pressure measurements will be collected in millimeter of mercury (mmHg) and findings will be summarized using descriptive statistics including mean values and change from baseline values, as well as numbers of subjects with values outside limits of the normal range at each time point.
Assessment of safety by measuring vital signs - pulse | 12 Weeks
  Participant heart rate will be collected at screening, randomization and end of participation (Week 12 or early termination). Heart rate will be measured in beats per minute (bpm) and findings will be summarized using descriptive statistics including mean values and change from baseline values, as well as numbers of subjects with values outside limits of the normal range at each time point.
Assessment of safety through collection of concomitant medication usage information | 12 Weeks
  Use of concomitant medications and related information will be collected from time of ICF signing through end of participation (Week 12 or early termination). Concomitant medications will be coded using the World Health Organization (WHO) Drug Dictionary (WHODrug) and summarized by drug class with subject counts and percent.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Manley, Study Chair — Paratek Pharma
Locations (21):
- United States (21):
  - San Tan Allergy & Asthma, Gilbert, Arizona
  - Children's Hospital of Orange County, Orange, California
  - DaVinci Research, LLC, Sacramento, California
  - Breathe Clear Institute, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Colorado ENT & Allergy, Colorado Springs, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Kentuckiana ENT, Louisville, Kentucky
  - Centers for Advanced ENT Care, Towson, Maryland
  - University of Missouri Medical Center, Columbia, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - Allergy, Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, Tulsa, Oklahoma
  - Charleston ENT & Allergy, North Charleston, South Carolina
  - Carolina ENT Clinic/CENTRI Inc., Orangeburg, South Carolina
  - Orion Clinical Research, Austin, Texas
  - STAAMP Research, San Antonio, Texas
  - Alamo ENT Associates, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - EVMS at Old Dominion University, Norfolk, Virginia